CLINICAL TRIAL: NCT03743909
Title: Expression of Aberrant CD Markers in Acute Leukemia:Retrospective Study in South Egypt Cancer Institute
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mervat Awad Mohamed Ibrahim, South Egypt cancer institute Assuit university, Assiut University
Other Study IDs: acute leukemia
Record Dates: First submitted 2018-11-14; First posted 2018-11-16 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Acute Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with aberrant CD markers: by flowcytometry from hospital information system
- patients without aberrant CD markers: by flowcytometry from hospital information system

SUMMARY:
* To determine incidence of Expression of aberrant CD markers in acute leukemia in South Egypt .
* Correlation between this expression and outcome of the patient.

DETAILED DESCRIPTION:
"Acute leukemia" is defined by the World Health organization standards, in which greater than 20% of the cells in the bone marrow are blasts (Kabuto et al., 2006).

Acute leukemia is a cloned expansion of tumor cells in bone marrow, blood or other tissues. The acute leukemia is classified as acute myeloid leukemia (AML) due to defective differentiation of myeloid lineage or acute lymphoid leukemia (ALL) due to defective differentiation of lymphoid lineage(Olaniyi JA et al., 2011).

Leukemia is diagnosed by morphology and cytochemical examination of blast cells, immunophenotyping, cytogenetic and molecular genetics. (Hazarika M et al., 2015 ). immunophenotyping is mandatory for the diagnosis of hematolymphoid malignancies (Craig FE et al., 2008)

Immunophenotyping of leukemia cells plays crucial role in identification of leukemia cell line, assesment of maturation stage and finding possible aberrant antigens which in turn serves for individual treatment monitoring and detection of residual disease(Kahng J et al.,2008).

Immunophenotyping identifies cell surface/CD markers(cluster of differentiation), expressed at different stages of cell development, by applying monoclonal antibodies against them helps in the diagnosis and classification of leukemia. The morphologically similar blast cells can be easily differentiated by immunophenotyping on the basis of expression and different CD markers (Angelescu S et al.,2012).

Aberrant expression of CD markers has been observed in several cases of acute leukemia(Chang Y et al., 2011).

Aberrant phenotype is a phenomenon in which lymphoid-associated and other myeloid lineage markers expressed in myeloblasts or myeloid-associated markers expressed in lymphoblasts. Aberrant phenotype incidence has been reported in both ALL and AML with varying frequencies as high as 88%(Macedo A et al.,1995).

The aberrant phenotypes are classified into different types: co-expression of lymphoid-associated antigens or lineage infidelity; asynchronous antigen expression, in which early antigens are coexpressed with more mature ones; or antigen overexpression and existence of abnormal light scatter patterns(Gert Ossenkoppele et al., 2011).

Presence or absence of these aberrant markers may also be associated with poor or favorable prognosis(Alhan C et al., 2014).

Several studies have reported correlations of aberrantly expressed markers with clinical outcome in AML. For example, CD7 and CD25 expression has been associated with poor prognosis in normal karyotype AML(Cerny J et al.,2013) The IL3 receptor alfa (CD123) is overexpressed in 45% of AML patients, and this higher expression has also been associated with poor outcome (Riccioni R et al.,2002).

CD13 and CD33 are most frequently associated with aberrant myeloid expression in ALL (Hrusák O et al,2002).Studies indicate that aberrant immunophenotypic expression can decrease the time of remission and survival in children with ALL (Kurec et al., 1991).Aberrant expression of CD13 in ≥ 5% of blasts of adult patients with ALL is an adverse prognostic factor,that should be considered for more aggressive treatment(Dalal BI1 et al.,2014).

ELIGIBILITY:
Inclusion Criteria:

* All cases of acute leukemia in South Egypt Cancer Institute.

Exclusion Criteria:

* Cases outside South Egypt Cancer Institute.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: acute leukemia patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Expression of aberrant CD markers in acute leukemia by flowcytometry : Retrospective study in South Egypt Cancer Institute | 2008-2018
  * To determine incidence of Expression of aberrant CD markers in acute leukemia in South Egypt .
  * Correlation between this expression and outcome of the patient.